CLINICAL TRIAL: NCT00919100
Title: Buzzy: An Integration of Vibration, Cold, and Distraction for Pediatric Needle Pain Relief
Brief Title: Buzzy Versus Vapocoolant Spray: Pediatric Needle Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Principal Investigator, Lindsey L Cohen, PhD, Principal Investigator, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CON007573
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Pain
Keywords: pediatric; venipuncture; pain; vibration; vapocoolant
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Care (Other): venipuncture with vapocoolant spray offered
  Interventions: Other: vapocoolant
- Buzzy (Experimental): Vibrating device with cold pack held to arm with tourniquet proximal to venipuncture site, optional distraction cards.
  Interventions: Device: Buzzy

INTERVENTIONS:
Device: Buzzy — "Buzzy" is a vibrating cold pack attached with Velcro strap or tourniquet 5-10cm proximal to the site of venipuncture. The vibration is activated and the device remains in place throughout the procedure. The distraction cards are offered to the parents to show the children, with questions on the back and pictures on the front.
  Other Names: BuzzyR
  Arms: Buzzy
Other: vapocoolant — venipuncture with vapocoolant spray offered
  Other Names: PainEase
  Arms: Standard Care

SUMMARY:
A vibrating cold pack placed proximal to the site of venipuncture will decrease the pain of cannulation when compared to vapocoolant spray.

DETAILED DESCRIPTION:
Needle pain is the most common and the most feared source of childhood pain, resulting in needle phobia for 10% of adults. Current pain relief options include numbing creams, vapocoolant spray, or injected lidocaine. 17 million pediatric IV access procedures are done yearly with no pain intervention. An inexpensive, immediately acting form of needle pain control could reduce needle phobia in the long term if demonstrated to be effective for needle pain.

This study will evaluate pain self report and parent report using the Faces Pain Scale revised, and video-coded OSBD-R scores for patients undergoing emergency department venous access or cannulation procedures. Demographic information, pre-procedural anxiety, and success data from the attempts at placement will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring venipuncture in a pediatric emergency department
* Informed consent
* Patient assent

Exclusion criteria:

* Patients with sickle cell or other sensitivity to cold
* Nerve damage in the area
* Abrasion or break in skin where device would be placed
* Critically ill

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Baxter, MD, Principal Investigator — Children's Healthcare of Atlanta; Lindsey L Cohen, PhD, Principal Investigator — Georgia State University
Locations (1):
- Children's Healthcare of Atlanta, Scottish Rite, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Willing to share deidentified data with anyone interested in similar research.

REFERENCES:
- [Derived] Baxter AL, Cohen LL, McElvery HL, Lawson ML, von Baeyer CL. An integration of vibration and cold relieves venipuncture pain in a pediatric emergency department. Pediatr Emerg Care. 2011 Dec;27(12):1151-6. doi: 10.1097/PEC.0b013e318237ace4. PMID 22134226

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Buzzy
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Buzzy | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 41 | 81
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 9.91 [6.68 to 11.08] | 10.10 [8.91 to 11.99] | 10.0 [6.68 to 11.99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 18 | 25 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Faces Pain Scale-Revised (FPS-R)
Description: Self-report measure of pain via 6 faces ranging from neutral to increasing pain expression. The scoring for the scale ranges from 0-10 with lower scores representing lower pain and higher scores representing higher pain. The FPS-R was conducted several minutes following venipuncture. This time was not tracked, but it was typically between 2-5 minutes following completion of the venipuncture.
Time Frame: 5 minute
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Standard Care | Buzzy
Number analyzed (Participants) | 40 | 41
units on a scale | 4 [2 to 6] | 2 [2 to 2]

2. Secondary Outcome: OSBD-R Observational Pain/Distress Scale
Description: The Observational Scale of Behavioral Distress (OSBD) is a validated and commonly used scale. There are 11 OSBD distress responses (information seeking, cry, scream, physical restraint, verbal resistance, seeking emotional support, verbal pain, flail, verbal fear, muscular rigidity, and nervous behavior). Using videotapes of the venipuncture, a composite OSBD score of 1 (low distress) to 11 (high distress) was assigned from the time of placement of tourniquet to placement of the bandage or securing the intravenous line (IV) after the first attempt. Two students not associated with the hospital or the device had been previously trained in this methodology and coded all tapes. A supervisor assessed interrater reliability on each coded behavior. After each group of 10 subjects, interrater agreements that fell below the level of excellent agreement (kappa = 0.80) were reviewed and discussed by both coders, with the consensus score recorded and definitions of observed behaviors.
Time Frame: 5 minute
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Standard Care | Buzzy
Number analyzed (Participants) | 40 | 41
units on a scale | 2 [1 to 3] | 1 [0 to 2]

3. Secondary Outcome: Number of Participants With Venipuncture Success in One Attempt
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Buzzy
Number analyzed (Participants) | 40 | 41
Participants | 26 | 35

ADVERSE EVENTS:
Arm/Group | Standard Care | Buzzy
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No